CLINICAL TRIAL: NCT00684671
Title: Challenge Dose Administration of Twinrix™ or Comparator 4 Years After Primary Vaccination.
Brief Title: Evaluation of Immune Memory to Twinrix or Comparator by Challenge Dose Administration 4 Years After Primary Vaccination
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 111572
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Results first posted 2009-12-03 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis A; Hepatitis B
Keywords: Immune memory; Combined hepatitis A and B vaccine; > 41 years old
MeSH Terms: conditions — Hepatitis A; Hepatitis B | interventions — twinrix; Engerix-B; Hepatitis A Vaccines; Hepatitis B Vaccines

ARMS (3):
- Twinrix Group (Experimental): Subjects received a single challenge dose of combined hepatitis A/hepatitis B vaccine (Twinrix).
  Interventions: Biological: Twinrix
- Engerix + Havrix Group (Active Comparator): Subjects received separate administration of a single challenge dose of hepatitis B vaccine (Engerix) and hepatitis A vaccine (Havrix).
  Interventions: Biological: Engerix-B; Biological: Havrix
- HB VAX PRO + Vaqta Group (Active Comparator): Subjects received separate administration of a single challenge dose of hepatitis B vaccine (HB VAX PRO) and hepatitis A vaccine (Vaqta).
  Interventions: Biological: HBVAXPRO; Biological: Vaqta

INTERVENTIONS:
Biological: Twinrix — Intramuscular injection, single dose in left deltoid.
  Arms: Twinrix Group
Biological: Engerix-B — Intramuscular injection, single dose in left deltoid.
  Arms: Engerix + Havrix Group
Biological: Havrix — Intramuscular injection, single dose in right deltoid.
  Arms: Engerix + Havrix Group
Biological: HBVAXPRO — Intramuscular injection, single dose in the left deltoid.
  Arms: HB VAX PRO + Vaqta Group
Biological: Vaqta — Intramuscular injection, single dose in right deltoid.
  Arms: HB VAX PRO + Vaqta Group

SUMMARY:
Only subjects who participated in the primary study will be invited to participate in the extension phase and the challenge dose phase of this study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol.
* A male or female who completed the primary vaccination phase of the HAB-160 study (NCT 00603252).
* Written informed consent obtained from the subject.
* If the subject is female, she must be of non-childbearing potential; or, if of childbearing potential, she must be abstinent or have used adequate contraceptive precautions for 30 days prior to vaccination, have a negative pregnancy test and must agree to continue such precautions for two months after the vaccination.

Exclusion Criteria:

The following criteria should be checked at the time of study entry. If any apply, the subject must not be included in the study:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines within 30 days preceding the challenge dose, or planned use during the study period.
* History of any hepatitis A or hepatitis B vaccination or infection since the primary vaccination study.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Acute disease at the time of enrolment.
* Pregnant or lactating female.

Min Age: 41 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 506 (Actual)
Dates: Start 2008-05-26; Primary Completion 2008-11-03 (Actual); Study Completion 2008-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Wilrijk, Belgium
- GSK Investigational Site, Hradec Králové, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Chlibek R, von Sonnenburg F, Van Damme P, Smetana J, Tichy P, Gunapalaiah B, Leyssen M, Jacquet JM. Antibody persistence and immune memory 4 years post-vaccination with combined hepatitis A and B vaccine in adults aged over 40 years. J Travel Med. 2011 Mar-Apr;18(2):145-8. doi: 10.1111/j.1708-8305.2010.00499.x. Epub 2011 Feb 7. PMID 21366801
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 111572 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111572 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111572 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111572 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111572 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111572 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Twinrix Group | Engerix + Havrix Group | HB VAX PRO + Vaqta Group
Started | 172 | 170 | 164
Completed | 169 | 170 | 164
Not Completed | 3 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Alcoholic dependance | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Twinrix Group | Engerix + Havrix Group | HB VAX PRO + Vaqta Group | Total
Number analyzed (Participants) | 172 | 170 | 164 | 506
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (8.70) | 59.5 (10.18) | 59.1 (9.16) | 59.0 (9.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 83 | 85 | 253
  Male | 87 | 87 | 79 | 253

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Anamnestic Response to the Challenge Dose for Anti-hepatitis A (Anti-HAV) Antibodies
Description: Anamnestic response was defined as:
  * for initially seronegative subjects, antibody concentration greater than or equal the cut-off [≥ 15 Milli-International Units per Milliliter (mIU/mL)],
  * for initially seropositive subjects with pre-vaccination antibody, concentration < 100 mIU/mL: antibody concentration at least four times the pre-vaccination antibody concentration,
  * for initially seropositive subjects with pre-vaccination antibody concentration ≥ 100 mIU/mL: antibody concentration at least two times the pre-vaccination antibody concentration.
Time Frame: One month after the challenge dose.
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for analysis of immunogenicity.
Measure: Count of Participants; unit: Participants
Arm/Group | Twinrix Group | Engerix + Havrix Group | HB VAX PRO + Vaqta Group
Number analyzed (Participants) | 167 | 168 | 163
Participants | 164 | 164 | 162

2. Primary Outcome: Number of Subjects With Anamnestic Response to the Challenge Dose for Anti-hepatitis B Surface Antigen (Anti-HBs) Antibodies
Description: Anamnestic response was defined as :
  * for initially seronegative subjects, antibody concentration ≥ 10 Milli-International Units per Milliliter (mIU/mL),
  * for initially seropositive subjects: antibody concentration at ≥ 4 fold the pre-vaccination antibody concentration.
Time Frame: One month after the challenge dose.
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for analysis of immunogenicity.
Measure: Count of Participants; unit: Participants
Arm/Group | Twinrix Group | Engerix + Havrix Group | HB VAX PRO + Vaqta Group
Number analyzed (Participants) | 167 | 168 | 163
Participants | 156 | 148 | 136

3. Secondary Outcome: Anti-hepatitis A (Anti-HAV) and Anti-hepatitis B Surface Antigen (Anti-HBs) Antibody Concentrations
Description: Concentrations are given as geometric mean concentration (GMCs) expressed as mIU/mL.
Time Frame: Prior to administration of challenge dose
Population: Analysis was performed on the Long-Term According-to-Protocol (LT ATP) cohort for analysis of immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Twinrix Group | Engerix + Havrix Group | HB VAX PRO + Vaqta Group
Number analyzed (Participants) | 167 | 168 | 163
mIU/mL
  anti-HAV | 212.2 [177.5 to 253.7] | 175.4 [147.3 to 208.9] | 308.4 [255.6 to 372.1]
  anti-HBs | 40.3 [30.0 to 54.2] | 26.7 [19.6 to 36.3] | 15.4 [12.2 to 19.5]

4. Secondary Outcome: Anti-hepatitis A (Anti-HAV) and Anti-hepatitis B Surface Antigen (Anti-HBs) Antibody Concentrations
Description: Concentrations are given as geometric mean concentration (GMCs) expressed as mIU/mL.
Time Frame: Two weeks and one month after the challenge dose
Population: Analysis was performed on the Log-Term According-to-Protocol (LT ATP) cohort for analysis of immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Twinrix Group | Engerix + Havrix Group | HB VAX PRO + Vaqta Group
Number analyzed (Participants) | 167 | 168 | 163
mIU/mL
  Anti-HAV (at Day 14) | 2255.0 [2255.0 to 2636.8] | 1774.3 [1493.5 to 2107.9] | 2712.9 [2290.4 to 3213.3]
  Anti-HAV (at Day 30) | 4062.0 [3451.1 to 4781.0] | 3124.1 [2630.4 to 3710.5] | 7481.6 [6358.3 to 8803.3]
  Anti-HBs (at Day 14) | 8936.9 [6071.1 to 13155.4] | 1521.0 [1012.5 to 2285.0] | 1222.4 [821.3 to 1819.3]
  Anti-HBs (at Day 30) | 7233.7 [4868.2 to 10748.7] | 1242.5 [823.5 to 1874.8] | 1075.1 [717.2 to 1611.4]

5. Secondary Outcome: Number of Subjects Reporting Solicited Symptoms
Description: Solicited local symptoms assessed include pain, redness and swelling. Solicited general symptoms assessed include fatigue, gastrointestinal symptoms, headache and temperature (above 37 degree Celsius).
Time Frame: During the 4-day follow-up period after the challenge dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Twinrix Group | Engerix + Havrix Group | HB VAX PRO + Vaqta Group
Number analyzed (Participants) | 172 | 170 | 164
Participants
  Pain | 42 | 35 | 46
  Redness | 22 | 10 | 19
  Swelling | 9 | 3 | 12
  Fatigue | 29 | 24 | 28
  Gastrointestinal symptoms | 5 | 8 | 5
  Headache | 21 | 20 | 18
  Temperature | 2 | 0 | 2

6. Secondary Outcome: Number of Subjects Reporting Unsolicited Symptoms
Description: Unsolicited symptoms = any adverse event (AE) reported in addition to those solicited during the clinical study. Also any "solicited" symptom with onset outside the specified period of follow-up for solicited symptoms was reported as an unsolicited adverse event.
Time Frame: During the 31-day follow-up period after the challenge dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Twinrix Group | Engerix + Havrix Group | HB VAX PRO + Vaqta Group
Number analyzed (Participants) | 172 | 170 | 164
Participants | 28 | 10 | 21

7. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs) Since the Last Study Visit of the HAB-160 (NCT00603252) Long-term Follow-up Study Considered by the Investigator to Have a Causal Relationship to Primary Vaccination
Description: A serious adverse event (SAE) is any untoward medical occurrence that results in death, is life-threatening, requires hospitalisation or prolongation of existing hospitalisation, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study subject, or is a sign of suspected or confirmed hepatitis A or hepatitis B.
Time Frame: Since the last study visit of the primary study long-term follow-up study up to challenge dose administration (1 year)
Measure: Count of Participants; unit: Participants
Arm/Group | Twinrix Group | Engerix + Havrix Group | HB VAX PRO + Vaqta Group
Number analyzed (Participants) | 172 | 170 | 164
Participants | 0 | 0 | 0

8. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: as for outcome 7
Time Frame: During one month following the administration of the challenge dose
Measure: Count of Participants; unit: Participants
Arm/Group | Twinrix Group | Engerix + Havrix Group | HB VAX PRO + Vaqta Group
Number analyzed (Participants) | 172 | 170 | 164
Participants | 1 | 2 | 0

ADVERSE EVENTS:
Arm/Group | Twinrix Group | Engerix + Havrix Group | HB VAX PRO + Vaqta Group
Serious Adverse Events (participants affected / at risk) | 1/172 | 2/170 | 0/164
Other Adverse Events (participants affected / at risk) | 76/172 | 57/170 | 75/164
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Twinrix Group (N=172) | Engerix + Havrix Group (N=170) | HB VAX PRO + Vaqta Group (N=164)
Arterial occlusive disease (Vascular disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Nephritis interstitial (Renal and urinary disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Twinrix Group (N=172) | Engerix + Havrix Group (N=170) | HB VAX PRO + Vaqta Group (N=164)
Pain (General disorders) | 42 | 35 | 46
Redness (General disorders) | 22 | 10 | 19
Swelling (General disorders) | 9 | 3 | 12
Fatigue (General disorders) | 29 | 24 | 28
Headache (General disorders) | 21 | 20 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.